CLINICAL TRIAL: NCT04234724
Title: Physiological Effects of ANGPTL3 Variants in Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 833684; R01HL148769 (NIH)
Record Dates: First submitted 2019-12-04; First posted 2020-01-21 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hypocholesterolemia
Keywords: Angiopoietin-like protein 3 deficiency; Lipid Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Variant (Experimental): Volunteers with known ANGPTL3 variants
  Interventions: Other: Kinetics test, oral fat tolerance test, and an oral glucose tolerance test.
- Non-variant (Other): Healthy volunteers with no ANGPTL3 variants
  Interventions: Other: Kinetics test, oral fat tolerance test, and an oral glucose tolerance test.

INTERVENTIONS:
Other: Kinetics test, oral fat tolerance test, and an oral glucose tolerance test. — Subjects will participate in a kinetics test, oral fat tolerance test, and an oral glucose tolerance test.

SUMMARY:
To evaluate the role of ANGPTL3, on lipid metabolism. To explore the role of this protein on glucose metabolism.

DETAILED DESCRIPTION:
Oral fast tolerance test, lipoprotein kinetics and a glucose tolerance test to evaluate the role of ANGPTL3, on lipid metabolism and to explore the role of this protein on glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 or older meeting at least one of the following criteria

  1. Carrying genetic variants in the gene encoding for ANGPTL3,
  2. Unaffected controls matched for age, race, gender,
  3. Willing to follow study procedures
  4. Able to provide inform consent

     Exclusion Criteria:
* Any medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study, or confound the study data
* Taking any medication that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study, or confound the study data
* Women that are pregnant or nursing
* History of liver disease or abnormal liver function tests (>2x upper limit of normal)
* History of kidney disease or chronic renal insufficiency (eGFR <60 mL/min/1.73 m2)
* Uncontrolled hypertension (>160/100 mmHg)
* Uncontrolled diabetes
* Anemia (hemoglobin <11.0 mg/dL) History of a non-skin malignancy within the previous 5 years Major surgery within the past 3 months
* History of any organ transplant
* History of alcohol or drug abuse
* Participation in clinical trials assessing the efficacy and safety of drugs affecting lipid metabolism within the past 6 weeks (or longer depending on the known half-life of the drug) that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study, or confound the study data
* Inability to comply to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The role of ANGPTL3 on lipid metabolism. | through study completion, an average of 13 weeks
  Assessing ApoB-containing lipoprotein fractional catabolic rate
The role of this protein on glucose metabolism. | through study completion, an average of 13 weeks
  Looking for glucose area under the curve following Oral Glucose Tolerance Test
The role of ANPTL3 on fatty acids | through study completion, an average of 13 weeks
  Looking for fatty acids area under the curve following Oral Fat Tolerance Test

CONTACTS AND LOCATIONS:
Overall Officials: Marina Cuchel, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT04234724/ICF_000.pdf